CLINICAL TRIAL: NCT06359470
Title: 3D CT Scan of the Modified Reversed Contralateral Axial Rotation Position in Patients With Lumbar Disc Prolapse. A New Manual Nerve Decompression Position.
Brief Title: the Modified Reversed Contralateral Axial Rotation Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Noha Khaled Shoukry (Other)
Responsible Party: Sponsor-Investigator, Noha Khaled Shoukry, lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CaiUni
Record Dates: First submitted 2024-04-04; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Disc Prolapse With Radiculopathy

STUDY DESIGN:
Intervention Model Description: This study was conducted on ninety male patients (30 in each group), ages ranged from 20 - 40 years old, and were diagnosed with unilateral lumbar disc prolapse (group1: L3-L4), (group 2: L4- L5) and (group 3: L5-S1) for at least three months in a radiology center specialized in the spine (Egyscan center). Each group was imaged three times (from the supine position, then from the oblique position after 10 minutes, and finally from the oblique position again after 48 hours). The oblique image was taken during a specific trunk position the modified reversed contralateral rotation (side-lying with side bending to the non-affected side and rotation to non affected side).The CSA of LIVF and SLR test was assessed at the three times of testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- positioning (Experimental): the supine position, then from the oblique position after 10 minutes, and finally from the oblique position again after 48 hours
  Interventions: Other: Positioning technique

INTERVENTIONS:
Other: Positioning technique — First time of testing: Firstly, the patients were scanned in the conventional neutral supine position and a 3D-CT scan was taken.
  Second time of testing: after 10 minutes, the patients were scanned in the modified reversed contralateral rotation (side-lying on a hard pillow with side bending to the non-affected side and rotation to non affected side). This is achieved through instructing the participant to first lie on the side lying on a wedge pillow (that is flexible with dimensions of 30 cm in height and 75 cm in length) to achieve trunk side bending to non-affected side this pillow is the same for all patients, then the patient/participant rotated to the affected side (pelvis on the trunk rotation), and 3D-CT scan.
  Third time of testing: after 48 hours, the patients were scanned in the modified reversed contralateral rotation.

SUMMARY:
This study aimed to investigate the effect of specific three-dimensional (3D) positions of the trunk on patients with lumbar discogenic pain with radiculopathy aiming to find a position that directly decompresses the impinged root as well as the effect of this position on the CSA of the L3-L4, L4-L5 and L5-S1 intervertebral foramen (IVF) using 3D-CT scan imaging of the real spine

DETAILED DESCRIPTION:
Background: Management of lumbar discogenic pain is complex and there is ongoing debate over both surgical and conventional conservative treatments. Purpose: This study aimed to investigate the real-time effect of specific three-dimensional (3D) positions of the trunk on patients with lumbar discogenic pain with radiculopathy aiming to find a position that directly decompresses the impinged root as well as the effect of this position on the CSA of the L3-L4, L4-L5 and L5-S1 intervertebral foramen (IVF) using 3D-CT scan imaging of the real spine. Methods: This study was conducted on ninety male patients (30 in each group), ages ranged from 20 - 40 years old, and were diagnosed with unilateral lumbar disc prolapse (group1: L3-L4), (group 2: L4- L5) and (group 3: L5-S1) for at least three months in a radiology center specialized in the spine (Egyscan center). Each group was imaged three times (from the supine position, then from the oblique position after 10 minutes, and finally from the oblique position again after 48 hours). The oblique image was taken during a specific trunk position the modified reversed contralateral rotation (side-lying on a hard pillow with side bending to the non-affected side and rotation to non affected side).The CSA of LIVF and SLR test were assessed at the three times of testing Results: The mixed design MANOVA revealed that the mean values of the LIVF CSA and the SLR significantly increased in the reversed contralateral rotation position after 48 hours compared to the same position after 10 minutes and the supine position in the three tested groups (P=0.001). Moreover, the LIVF CSA and the SLR significantly increased in the reversed contralateral rotation position after 10 minutes compared to the supine position in the three tested groups (P=0.001). Conclusion: Modified reversed contralateral rotation of the trunk has a real-time decompressing effect on patients with lumbar disc prolapse as well as a significantly increasing effect on the CSA of L3-L4, L4-L5 and L5-S1 IVF in the three tested groups. Changing the spine position from supine to the modified reversed contralateral rotation position had a great clinical value on patients with lumbar discogenic pain with radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

* All patients had a second-grade disc bulge (2-3mm) which was detected from the T2 axial view of MRI. All patients had radiculopathy due to lumbar disc prolapse. The diagnosis was confirmed by physical, neurological examination (motor assessment, sensory assessment, reflexes), and radiological assessment (CT or MRI)

Exclusion Criteria:

* bilateral and multilevel disc prolapse, sequestrated , migrated and disc herniation defined by MRI , acute onset of pain (pain less than three months), presence of active infection in the lumbar spine, any spinal deformities e.g., moderate, or severe scoliosis deformity (Cobb angle ≥ 25°), postoperative cases, Cauda equine lesion, the presence of any comorbidities, history of patients who suffered from cancer, unexplained weight loss, immunosuppression, prolonged use of steroids, intravenous drug use, urinary tract infection, pain that is increased or unrelieved by rest, fever, significant trauma related to age, bladder or bowel incontinence, urinary retention (with overflow incontinence), saddle anesthesia, loss of anal sphincter tone, major motor weakness in lower extremities, fever, and vertebral tenderness

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-11-05 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-01-14 (Actual)

PRIMARY OUTCOMES:
Straight leg raising test | 48 hours
  With the patient in the supine position and the hips were neutral, neither abducted nor adducted nor rotated, the investigator lifted the leg slowly while the knee was kept in extended position. Each leg is raised separately until pain occurs. When the patient reported feeling radiating pain the angle between the bed and the leg was recorded by a goniometer

SECONDARY OUTCOMES:
Foraminal cross sectional area | 48 hours
  The foraminal area was defined as the outline of the LIVF. It is measured by the boundary of the adjacent superior and inferior vertebral pedicles, the posterosuperior portion of the inferior vertebral body, the posterior portion of the intervertebral disc, the posteroinferior portion of the superior vertebral body, and the anterior portion of ligamentum flavum

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No